CLINICAL TRIAL: NCT01148446
Title: A Randomized Phase III Randomized Study to Compare R-CHOP Versus R-mini-CEOP in Elderly Patients (>65 Years) With Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: R-CHOP Versus R-mini-CEOP in Elderly Patients(>65)With DLBCL
Acronym: ANZINTER3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Francesco Merli, MD, U.O.A. di Ematologia Azienda Ospedaliera S. Maria Nuova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIL ANZINTER3
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Elderly Patients (>65 Years); Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: DLBCL; R-CHOP; R-CEOP; Elderly patients
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Epirubicin; Vinblastine; Rituximab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-CHOP (Experimental): R-CHOP (every 21 days) for six courses Cyclophosphamide: 750 mg/m2, IV, day 1 Doxorubicin: 50 mg/m2, IV, day 1 Vincristine: 1.4 (max 2) mg/m2, IV, day 1 Prednisone: 75 mg/m2, IV, days 1-5 Rituximab: 375 mg/m2, IV, day 1 G-CSF: 300 µg tota, SC; days 7-11
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab; Drug: G-CSF
- R-mini-CEOP (Experimental): R-miniCEOP (every 21 days)for six courses Cyclophosphamide: 50 mg/m2, IV, day 1 Epirubicin: 50 mg/m2, IV, day 1 Vinblastine: 5 mg/m2, IV, day 1 Prednisone: 60 mg/m2, IV/PO, days 1-5 Rituximab: 375 mg/m2, IV, day 1 G-CSF: 300 µg tota, SC; days 7-11
  Interventions: Drug: Cyclophosphamide; Drug: Prednisone; Drug: Epirubicin; Drug: Vinblastine; Drug: Rituximab; Drug: G-CSF

INTERVENTIONS:
Drug: Cyclophosphamide — 750 mg/mq IV, day 1
  Arms: R-CHOP
Drug: Cyclophosphamide — 50 mg/mq IV, day 1
  Arms: R-mini-CEOP
Drug: Doxorubicin — 50 mg/mq IV, day1
  Arms: R-CHOP
Drug: Vincristine — 1,4 mg/mq (max 2 mg)IV, day 1
  Arms: R-CHOP
Drug: Prednisone — 75 mg/mq IV, days 1-5
  Arms: R-CHOP
Drug: Prednisone — 60 mg/mq IV/PO, days 1-5
  Arms: R-mini-CEOP
Drug: Epirubicin — 50 mg/mq IV, day 1
  Arms: R-mini-CEOP
Drug: Vinblastine — 5 mg/mq IV, day 1
  Arms: R-mini-CEOP
Drug: Rituximab — 375 mg/mq IV, day 1
Drug: G-CSF — 300 µg tot., SC; days 7-11

SUMMARY:
The study has the purpose to compare R-CHOP versus R-mini-CEOP in elderly patients (>65 years) with Diffuse Large B Cell Lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with untreated DLBCL aged 66 to 80 years without major accompanying diseases and considered as "non frail".
2. Patients were classified as "non frail" (fit) if they had

   * ADL (Activity of Daily Living) score of 6
   * less than three grade 3 Cumulative Illness Rating Score for Geriatrics (CIRS-G) co-morbidities and no grade 4 co-morbidities
   * absence of geriatric syndrome
3. Patients HIV negativity;
4. Concurrent malignancy;
5. Written Informed Consent.

Exclusion Criteria:

* All other patients were classified as "unfit", and were excluded from randomization

Ages: 66 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 226 (Actual)
Dates: Start 2003-01; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 2 years

SECONDARY OUTCOMES:
Complete Remission (CR) rate | 2 years
Disease Free Survival (DFS) | 2 years
Multidimensional Evaluation Scale for the definition of "frail" and "non frail" patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Merli, MD, Study Chair — U.O.A. di Ematologia Azienda Ospedale S. Maria Nuova; Marilena Bertini, MD, Study Chair — U.O.A. di Ematologia Ospedale Molinette
Locations (11):
- Italy (11):
  - S.C. di Ematologia, Spedali Civili, Brescia, Brescia
  - Ospedale di Vigevano, Vigevano, Pavia
  - Ospedale Garibaldi-Nesima, Catania
  - Ospedale civile Divisione di Ematologia, Civitanova Marche (MC)
  - Ospedale San Sebastiano, Correggio (RE)
  - Presidio Ospedaliero Annunziata, Cosenza
  - Istituto Vito Fazzi, Lecce
  - Azienda Ospedaliera Policlinico, Modena
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Ospedale civile DH oncologico, Sassuolo (MO)
  - Ospedale San Giovanni Battista - Molinette, Torino

REFERENCES:
- [Derived] Shi Q, Schmitz N, Ou FS, Dixon JG, Cunningham D, Pfreundschuh M, Seymour JF, Jaeger U, Habermann TM, Haioun C, Tilly H, Ghesquieres H, Merli F, Ziepert M, Herbrecht R, Flament J, Fu T, Coiffier B, Flowers CR. Progression-Free Survival as a Surrogate End Point for Overall Survival in First-Line Diffuse Large B-Cell Lymphoma: An Individual Patient-Level Analysis of Multiple Randomized Trials (SEAL). J Clin Oncol. 2018 Sep 1;36(25):2593-2602. doi: 10.1200/JCO.2018.77.9124. Epub 2018 Jul 5. PMID 29975624
- [Derived] Merli F, Luminari S, Rossi G, Mammi C, Marcheselli L, Tucci A, Ilariucci F, Chiappella A, Musso M, Di Rocco A, Stelitano C, Alvarez I, Baldini L, Mazza P, Salvi F, Arcari A, Fragasso A, Gobbi PG, Liberati AM, Federico M. Cyclophosphamide, doxorubicin, vincristine, prednisone and rituximab versus epirubicin, cyclophosphamide, vinblastine, prednisone and rituximab for the initial treatment of elderly "fit" patients with diffuse large B-cell lymphoma: results from the ANZINTER3 trial of the Intergruppo Italiano Linfomi. Leuk Lymphoma. 2012 Apr;53(4):581-8. doi: 10.3109/10428194.2011.621565. Epub 2011 Nov 15. PMID 21895543